CLINICAL TRIAL: NCT01167270
Title: The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) Study
Acronym: INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ian M. Paul, MD (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 34493; 1R01DK088244-01 (NIH)
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Infant; Obesity
Keywords: Infant Diet; Toddler Diet; Responsive Feeding; Infant Temperament; Parent competency; Childhood Obesity prevention; Rapid infant weight gain
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parenting Insight (Active Comparator): Educational program contains messages to provide developmentally appropriate guidance to parents of infants on responsive parenting and healthy lifestyle that will prevent rapid weight gain in infancy and overweight at age 3 years.
  Interventions: Behavioral: Parenting Insights
- Child Safety Insights (Placebo Comparator): A child safety intervention with messages focused on the infant's environment and interactions with parents. They will be guided by the AAP guidelines and the Academy's guide for health supervision, Bright Futures
  Interventions: Behavioral: Child Safety Insights

INTERVENTIONS:
Behavioral: Child Safety Insights — A child safety intervention with messages focused on the infant's environment and interactions with parents. They will be guided by the American Academy of Pediatrics as well as the Academy's guide for health supervision, Bright Futures.
  Arms: Child Safety Insights
Behavioral: Parenting Insights — Educational program contains messages to provide developmentally appropriate guidance to parents of infants on responsive parenting and healthy lifestyle that will prevent rapid weight gain in infancy and overweight at age 3 years.
  Arms: Parenting Insight

SUMMARY:
This study will test an intervention program designed to provide developmentally appropriate guidance to parents of infants on responsive parenting and healthy lifestyle to see if that intervention will prevent rapid weight gain in infancy and overweight at age 3 years. Further, compared with control infants, intervention infants will have lower body mass index (BMI) percentiles at age 3. The investigators also hypothesize that control infants will gain weight more rapidly over time.

DETAILED DESCRIPTION:
Principal Hypotheses: An intervention program designed to provide developmentally appropriate guidance to parents of infants on responsive parenting and healthy lifestyle will prevent rapid weight gain in infancy and overweight at age 3 years. Further, compared with control infants, intervention infants will have lower BMI percentiles at age 3. We also hypothesize that control infants will gain weight more rapidly over time, adjusting for trait-stable and time-varying covariates (e.g., maternal pre-pregnancy BMI, percent of feedings that are breast milk vs. formula, sleep duration, and feeding frequency).

The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) Study, will test these hypotheses in a two arm randomized trial where participants in a program to prevent childhood obesity will be compared with those in a child safety control program. Nurses will deliver interventions to first-time parents and their infants in both study groups at four home visits in the first year after birth followed by annual clinical research center visits until age 3. Blood samples for genetic testing on appetite, growth, and temperament will be collected from mother, child, and father. The obesity prevention program focuses on messages of responsive parenting and healthy lifestyle, extending from infancy through age 3 years. The intervention will teach first-time parents to interact with their infants in a way that is prompt, emotionally supportive, contingent, and developmentally appropriate. This information is especially important during the first year after birth as infants make a dramatic dietary transition from the initial exclusive milk diet to one with many foods of the adult diet of their culture. During this transition, as foods are being introduced to children, there are numerous opportunities to address dietary content as well as parent feeding style. In addition to these messages, intervention parents will be given education on growth charts, the meaning of growth chart percentiles, and healthy growth patterns during early life. The intervention program is hypothesized to show efficacy in both breast and formula fed infants as measured by the primary outcome, body mass index (BMI) percentile at age 3 years. Additionally, participants will be followed to collect anthropometric measurements at 4,5,6,10,14,and 17 years of age to provide significant insight into long-term obesity risk.

The proposed research adds two major pieces by enrolling second born siblings and collecting genetic specimens from both siblings and their parents. Specifically, this translational research will a) prospectively evaluate obesity-related parenting similarities and differences as well as weight-related outcomes between first and second-born siblings, b) explore how genetic differences among siblings that are associated with appetite, temperament, and obesity susceptibility affect parent-child interactions, degree of responsive parenting, and weight status, and c) determine whether INSIGHT study intervention carryover effects occur among families participating in the observation-only second-born child evaluation.

ELIGIBILITY:
Inclusion Criteria:

* full-term infant(> 37 0/7 weeks gestational age)discharged from hospital without significant morbidity
* singleton infant
* nursery/NICU/maternity stay of 7 days or less
* primiparous mother
* English speaking mother

Exclusion Criteria:

* presence of a congenital anomaly or neonatal condition that significantly affects a newborn's feeding (e.g. cleft lip, cleft palate, metabolic disease
* any major maternal morbidities and/or pre-existing condition that would affect postpartum care such as cancer, multiple sclerosis, lupus, etc.
* maternal age <=20 years
* prenatal ultrasound presence of intrauterine growth retardation (IUGR)
* infant birth weight <2500 grams plan for newborn to be adopted
* plan to move from Central Pennsylvania within 3 years
* inability to complete contact form with name, address, phone numbers, etc.
* Practicing pediatrician or pediatric resident

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-01; Primary Completion 2017-04 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
BMI percentile at 3 years | 3 years
  BMI percentile at 3 years

SECONDARY OUTCOMES:
Weight-for-length percentile at several intervals in the first 12 months after birth | 12 months of age
  Weight-for-length percentile at several intervals in the first 12 months after birth
BMI percentile at age 2 years | 2 years of age
  BMI percentile at age 2 years
Proportion of infants with BMI > 85th and 95th percentiles at ages 2 and 3 years | aged 2 and 3 years
  Proportion of infants with BMI > 85th and 95th percentiles at ages 2 and 3
Proportion of infants with accelerated weight gain between numerous study intervals | birth to 4 months, birth to 1 year, birth to 3 years, 1 year to 3 years
  Proportion of infants with accelerated weight gain between numerous study

OTHER OUTCOMES:
Factors that influence the succession of the oral and gut microbiomes. | birth to 1 year of age
  Microbiome samples collected from mother and baby throughout the first year of life (including stool and buccal swabs) are collected for analyses. Outcome only for the sibling study not the first born study

CONTACTS AND LOCATIONS:
Overall Officials: Leann L Birch, PhD, Principal Investigator — Penn State University; Ian M Paul, MD, MSc, Principal Investigator — Penn State College of Medicine and Children's Hospital
Locations (2):
- United States (2):
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Penn State University, State College, Pennsylvania

REFERENCES:
- [Background] Paul IM, Williams JS, Anzman-Frasca S, Beiler JS, Makova KD, Marini ME, Hess LB, Rzucidlo SE, Verdiglione N, Mindell JA, Birch LL. The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) study. BMC Pediatr. 2014 Jul 18;14:184. doi: 10.1186/1471-2431-14-184. PMID 25037579
- [Result] Paul IM, Savage JS, Anzman-Frasca S, Marini ME, Mindell JA, Birch LL. INSIGHT Responsive Parenting Intervention and Infant Sleep. Pediatrics. 2016 Jul;138(1):e20160762. doi: 10.1542/peds.2016-0762. PMID 27354460
- [Result] Savage JS, Birch LL, Marini M, Anzman-Frasca S, Paul IM. Effect of the INSIGHT Responsive Parenting Intervention on Rapid Infant Weight Gain and Overweight Status at Age 1 Year: A Randomized Clinical Trial. JAMA Pediatr. 2016 Aug 1;170(8):742-9. doi: 10.1001/jamapediatrics.2016.0445. PMID 27271455
- [Result] Paul IM, Hohman EE, Birch LL, Shelly A, Vallotton CD, Savage JS. Exploring infant signing to enhance responsive parenting: Findings from the INSIGHT study. Matern Child Nutr. 2019 Jul;15(3):e12800. doi: 10.1111/mcn.12800. Epub 2019 Mar 19. PMID 30810273
- [Result] Craig SJC, Blankenberg D, Parodi ACL, Paul IM, Birch LL, Savage JS, Marini ME, Stokes JL, Nekrutenko A, Reimherr M, Chiaromonte F, Makova KD. Child Weight Gain Trajectories Linked To Oral Microbiota Composition. Sci Rep. 2018 Sep 19;8(1):14030. doi: 10.1038/s41598-018-31866-9. PMID 30232389
- [Result] Eagleton SG, Hohman EE, Verdiglione N, Birch LL, Paul IM, Savage JS. INSIGHT Study Maternal Return to Work and Infant Weight Outcomes. Acad Pediatr. 2019 Jan-Feb;19(1):67-73. doi: 10.1016/j.acap.2018.08.008. Epub 2018 Aug 23. PMID 30145361
- [Result] Savage JS, Hohman EE, Marini ME, Shelly A, Paul IM, Birch LL. INSIGHT responsive parenting intervention and infant feeding practices: randomized clinical trial. Int J Behav Nutr Phys Act. 2018 Jul 9;15(1):64. doi: 10.1186/s12966-018-0700-6. PMID 29986721
- [Result] Paul IM, Savage JS, Anzman-Frasca S, Marini ME, Beiler JS, Hess LB, Loken E, Birch LL. Effect of a Responsive Parenting Educational Intervention on Childhood Weight Outcomes at 3 Years of Age: The INSIGHT Randomized Clinical Trial. JAMA. 2018 Aug 7;320(5):461-468. doi: 10.1001/jama.2018.9432. PMID 30088009
- [Result] Anzman-Frasca S, Paul IM, Moding KJ, Savage JS, Hohman EE, Birch LL. Effects of the INSIGHT Obesity Preventive Intervention on Reported and Observed Infant Temperament. J Dev Behav Pediatr. 2018 Dec;39(9):736-743. doi: 10.1097/DBP.0000000000000597. PMID 29927795
- [Result] Adams EL, Marini ME, Stokes J, Birch LL, Paul IM, Savage JS. INSIGHT responsive parenting intervention reduces infant's screen time and television exposure. Int J Behav Nutr Phys Act. 2018 Mar 15;15(1):24. doi: 10.1186/s12966-018-0657-5. PMID 29544506
- [Result] Hohman EE, Savage JS, Birch LL, Beiler JS, Paul IM. Pacifier Use and Early Life Weight Outcomes in the Intervention Nurses Start Infants Growing on Healthy Trajectories Study. Child Obes. 2018 Jan;14(1):58-66. doi: 10.1089/chi.2017.0177. Epub 2017 Oct 4. PMID 28976781
- [Result] Paul IM, Hohman EE, Loken E, Savage JS, Anzman-Frasca S, Carper P, Marini ME, Birch LL. Mother-Infant Room-Sharing and Sleep Outcomes in the INSIGHT Study. Pediatrics. 2017 Jul;140(1):e20170122. doi: 10.1542/peds.2017-0122. Epub 2017 Jun 5. PMID 28759407
- [Result] Carney MC, Tarasiuk A, DiAngelo SL, Silveyra P, Podany A, Birch LL, Paul IM, Kelleher S, Hicks SD. Metabolism-related microRNAs in maternal breast milk are influenced by premature delivery. Pediatr Res. 2017 Aug;82(2):226-236. doi: 10.1038/pr.2017.54. Epub 2017 May 24. PMID 28422941
- [Result] Hohman EE, Paul IM, Birch LL, Savage JS. INSIGHT responsive parenting intervention is associated with healthier patterns of dietary exposures in infants. Obesity (Silver Spring). 2017 Jan;25(1):185-191. doi: 10.1002/oby.21705. PMID 28008749
- [Derived] Dadzie A, Master L, Hohman EE, Acton EH, Tauriello S, Paul IM, Savage JS, Anzman-Frasca S, Buxton OM. Associations Between Sleep Health and Child Behavior at Age 6 Years in the INSIGHT Study. J Dev Behav Pediatr. 2025 Jan-Feb 01;46(1):e56-e63. doi: 10.1097/DBP.0000000000001326. Epub 2024 Nov 8. PMID 39514718
- [Derived] Hernandez Acton E, Kubiniec E, Bhargava S, Tauriello S, Paul IM, Savage JS, Anzman-Frasca S. INSIGHT responsive parenting intervention effects on child self-regulation at ages 3 and 6 years. Dev Psychol. 2025 Aug;61(8):1413-1426. doi: 10.1037/dev0001839. Epub 2024 Sep 26. PMID 39325391
- [Derived] Tauriello S, Savage JS, Goldsmith J, Kubiniec E, Paul IM, Anzman-Frasca S. Effect of the INSIGHT Responsive Parenting Intervention on Parenting and Child Behavior at Ages 3 and 6 Years. J Pediatr. 2023 Apr;255:72-79. doi: 10.1016/j.jpeds.2022.10.025. Epub 2022 Oct 29. PMID 37081779
- [Derived] Hohman EE, Savage JS, Marini ME, Anzman-Frasca S, Buxton OM, Loken E, Paul IM. Effect of the INSIGHT Firstborn Parenting Intervention on Secondborn Sleep. Pediatrics. 2022 Jul 1;150(1):e2021055244. doi: 10.1542/peds.2021-055244. PMID 35703026
- [Derived] Hyczko AV, Ruggiero CF, Hohman EE, Anzman-Frasca S, Savage JS, Birch LL, Paul IM. Sex Differences in Maternal Restrictive Feeding Practices in the Intervention Nurses Start Infants Growing on Healthy Trajectories Study. Acad Pediatr. 2021 Aug;21(6):1070-1076. doi: 10.1016/j.acap.2021.05.002. Epub 2021 May 19. PMID 34020105
- [Derived] Hohman EE, Savage JS, Birch LL, Paul IM. The Intervention Nurses Start Infants Growing on Healthy Trajectories (INSIGHT) Responsive Parenting Intervention for Firstborns Affects Dietary Intake of Secondborn Infants. J Nutr. 2020 Aug 1;150(8):2139-2146. doi: 10.1093/jn/nxaa135. PMID 32412629
- [Derived] Adams EL, Marini ME, Brick TR, Paul IM, Birch LL, Savage JS. Ecological momentary assessment of using food to soothe during infancy in the INSIGHT trial. Int J Behav Nutr Phys Act. 2019 Sep 5;16(1):79. doi: 10.1186/s12966-019-0837-y. PMID 31488156